CLINICAL TRIAL: NCT00302458
Title: A Double-blind, Randomized, Placebo-controlled, Crossover Study of Repeat Dosing of OROS® Methylphenidate Hydrochloride (CONCERTA®) and Immediate Release Methylphenidate Hydrochloride in Healthy Adults
Brief Title: A Study of Repeat Dosing of OROS® Methylphenidate Hydrochloride (CONCERTA®) and Immediate Release Methylphenidate Hydrochloride in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Assistant Director of the Clinical and Research Program in Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2005-P-001812
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- OROS-MPH + OROS-MPH (Experimental): OROS-Methylphenidate Will be administered during the first part of the day, and again during the separate part of the day.
  Interventions: Drug: OROS-Methylphenidate
- IR MPH + IR MPH (Experimental): Immediate release methylphenidate will be administered in the first part of the day followed by Immediate release methylphenidate in the second part of the day.
  Interventions: Drug: Immediate Release Methylphenidate
- Plabebo + Placebo (Placebo Comparator): Placebo will be administered during the first part of the day, and again during the second part of the day.
  Interventions: Drug: Placebo
- OROS MPH+ IR MPH (Experimental): Concerta will be administered in the first part of the day, followed by Immediate Release Methylphenidate in the second part of the day.
  Interventions: Drug: OROS-Methylphenidate; Drug: Immediate Release Methylphenidate
- IR MPH + OROS MPH (Experimental): Immediate release Methylphenidate will be administered in the first part of the day, followed by Concerta in the second part of the day
  Interventions: Drug: OROS-Methylphenidate; Drug: Immediate Release Methylphenidate

INTERVENTIONS:
Drug: OROS-Methylphenidate — Each dose of OROS MPH will be 72 mg which will be supplied as two 36 mg overencapsulated capsules
  Other Names: Concerta; OROS MPH
  Arms: IR MPH + OROS MPH; OROS MPH+ IR MPH; OROS-MPH + OROS-MPH
Drug: Immediate Release Methylphenidate — Each dose of IR MPH will be 40 mg which will be supplied as two 20 mg overencapsulated capsules
  Other Names: IR MPH; Ritalin
  Arms: IR MPH + IR MPH; IR MPH + OROS MPH; OROS MPH+ IR MPH
Drug: Placebo — Placebo will be administered during the first part of the day, and again during the second part of the day.
  Arms: Plabebo + Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, five-period crossover study to examine the likability of a repeated administration of immediate release methylphenidate hydrochloride (IR-MPH 40 mg) and OROS®-MPH (CONCERTA® 72 mg) in healthy adults. Hypotheses are as follows:

* Hypothesis 1: the subjective feelings of detection and likeability will be greater for periods of IR-MPH administration than after OROS-MPH administration irregardless of sequence;
* Hypothesis 2: the greater ratings of feelings of detection and likeability will be associated with the periods of most rapid change in plasma d-MPH and not with the magnitude of plasma d-MPH concentration (other than the OROS-MPH to IR-MPH condition in which they coincide), and
* Hypothesis 3: the subjective feelings of dislike will be greatest for the two conditions in which IR-MPH is the second condition.

DETAILED DESCRIPTION:
The main goal of this study is to assess whether the abuse liability potential of delayed, repeated administrations of different formulations of MPH is moderated by the oral delivery system in which a delivery system with slower onset may be safer than one with more rapid early release. To this end, the investigators will compare repeated administration of orally administered, therapeutic doses of a short (IR-MPH) and a long-acting formulation of MPH (OROS-MPH) in the following areas:

1. pharmacokinetic profile of MPH assessing rate of onset of MPH action (indexed through change in plasma level) and
2. abuse liability (indexed through detection and likeability).

The investigators will test all combinations of initial administration and then delayed (repeated) administration of the two formulations: IR-MPH to IR-MPH; IR-MPH to OROS-MPH; OROS-MPH to IR-MPH; OROS-MPH to OROS-MPH, and placebo to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females. With the exception of women who have been post-menopausal for a minimum of 12 months prior to screening and those who have undergone hysterectomy or bilateral oophorectomy, all female subjects must have a negative urine pregnancy test at both screening and at each admission to the research unit. All male and female subjects must have used a medically acceptable form of birth control for at least one month prior to screening and be willing to continue use during the study. Medically acceptable forms of birth control include abstinence, hormonal contraceptives, diaphragm with spermicide, condom with spermicide, intrauterine device, or surgical sterilization (including vasectomy of male partner[s]).
2. Eighteen (18) to 45 years of age, inclusive
3. Based on medical history, limited physical examination (neurologic and cardiac) and/or lab results, are considered healthy and free of any conditions that may interfere with participation in the study. Any abnormalities at screening on results of electrocardiogram (ECG) or any laboratory test must be determined to be not clinically significant by an investigator.
4. Agree to not use prescription stimulants (except for the study medication) during the study
5. Have venous access sufficient for blood sampling as determined by clinical examination
6. Weigh at least 100 pounds at screening
7. Agree and are available to return to the study center for five full-day (approximately 18 hours) study visits held five to 30 days apart within a 22-week period, and willing to complete all protocol-specified assessments.
8. Able to read and comprehend English

Exclusion Criteria:

1. Marked anxiety, tension, and agitation since the drug may aggravate these symptoms
2. Known hypersensitivity to methylphenidate or other components of Concerta or Ritalin
3. Subjects with glaucoma
4. Motor tics or with a family history or diagnosis of Tourette's syndrome
5. Treated with monoamine oxidase inhibitors (MAOIs) or within 14 days of discontinuation of treatment with MAOIs
6. Presence or history of any medically diagnosed, clinically significant Axis I psychiatric disorder (including substance use disorders, bipolar disorder, any psychotic disorder)
7. Scores of Baseline Scales:

   * Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale) (Hamilton 1960)
   * Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale) (Beck et al 1961)
   * Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) (Hamilton 1959)
8. Any clinically significant chronic disease or unstable medical abnormality by history or physical examination, including hypertension, hyperthyroidism, a seizure disorder, history of myocardial infarction or stroke, or history of cardiac arrhythmia or heart murmur (other than uncomplicated mitral valve prolapse)
9. Clinically significant abnormal baseline laboratory values which include the following:

   * Values > 20% above the upper range of the laboratory standard of a basic metabolic screen and complete blood count
   * Exclusionary blood pressure > 140 (systolic) and 90 (diastolic).
   * Exclusionary ECG parameters: QTC > 460 msec, QRS > 120 msec, and PR > 200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist
10. Currently taking or require any of the following medications:

    * Clonidine or other alpha-2 adrenergic receptor agonists
    * Tricyclic antidepressants
    * Selective serotonin reuptake inhibitors (SSRIs)
    * Theophylline
    * Coumarin anticoagulants
    * Anticonvulsants
    * Prescription stimulants
11. Have taken an SSRI in the 35 days before initiation of the study medication
12. Currently physically dependent on benzodiazepines, opiates or alcohol as determined by clinical evaluation or positive urine drug screen at screening
13. Preexisting severe gastrointestinal narrowing (pathologic or iatrogenic, for example: small bowel inflammatory disease, "short gut" syndrome due to adhesions or decreased transit time, past history of peritonitis, cystic fibrosis, chronic intestinal pseudoabsorption, or Meckel's diverticulum)
14. Unable to swallow the study medication whole
15. Have had a significant blood loss (> 500 mL) or donated blood in the 30 days preceding dosing
16. Have a positive urine drug screen at screening
17. Have taken an investigational medication or product within the past 30 days
18. Have taken prescription medications (with the exception of birth control methods) within seven days of screening or is anticipated to need any medications, over-the-counter products (other than acetaminophen), or herbal supplements during the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Spencer TJ, Biederman J, Martin JM, Moorehead TM, Mirto T, Clarke A, Batchelder H, Faraone SV. Importance of pharmacokinetic profile and timing of coadministration of short- and long-acting formulations of methylphenidate on patterns of subjective responses and abuse potential. Postgrad Med. 2012 Jan;124(1):166-73. doi: 10.3810/pgm.2012.01.2529. PMID 22314126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 2005 to 2007 at Massachusetts General Hospital and were recruited using IRB approved postings through web and email.
Pre-assignment Details: Based on a comprehensive screening, subjects who did not meet eligibility criteria for the study were excluded. Others withdrew or were lost to follow-up before randomization.
Groups:
- Healthy Volunteers: Healthy volunteers each received IR MPH, Oros MPH, and matched placebo (at four separate study visits) in a four way crossover design.
Period: Overall Study
Arm/Group | Healthy Volunteers
Started | 29
Completed | 26
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Ineligible after screening | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: One subject was ineligible, one subject was lost to follow-up, one withdrew, and twenty six subjects completed the study.
Groups:
- Healthy Volunteers: Healthy volunteers each received IR-MPH, OROS-MPH, and matched placebo (in four separate visits) in a four way crossover design.
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.86 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of d-Methylphenidate
Description: Objective measure determined from blood samples, measured 4 hours after the dose
Time Frame: 4 hours
Population: All subjects received each combination of medications on a separate day (total= 5 days)
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Placebo- Placebo: Healthy volunteers received a placebo, followed by a placebo four hours later
- IR-MPH + OROS MPH: Healthy volunteers received a dose of Immediatate Release Methylphenidate at hour 0, followed by a dose of OROS-Methylphenidate four hours later
- IR-MPH +IR-MPH: Healthy volunteers received a dose of Immediatate Release Methylphenidate at hour 0, followed by a dose of Immediate Release Methylphenidate four hours later
- OROS-MPH+OROS-MPH: Healthy volunteers received a dose of OROS-Methylphenidate at hour 0, followed by a dose of OROS-Methylphenidate four hours later
- OROS-MPH+ IR-MPH: Healthy volunteers received a dose of OROS-Methylphenidate at hour 0, followed by a dose of Immediate Release Methylphenidate four hours later
Arm/Group | Placebo- Placebo | IR-MPH + OROS MPH | IR-MPH +IR-MPH | OROS-MPH+OROS-MPH | OROS-MPH+ IR-MPH
Number analyzed (Participants) | 26 | 26 | 26 | 26 | 26
mg/L | 0.00 (0.00) | 15.06 (5.0) | 25.34 (7.3) | 20.34 (6.4) | 28.79 (8.3)

ADVERSE EVENTS:
Arm/Group | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteers (N=29)
Anxiety (Psychiatric disorders) | 7 (12)
Appetite Loss (Metabolism and nutrition disorders) | 14 (27)
Aware of heartbeat (Cardiac disorders) | 3 (4)
Chest Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Ear and labyrinth disorders) | 7 (8)
Dry Mouth (General disorders) | 12 (27)
Fatigue (General disorders) | 4 (7)
Flushing (General disorders) | 4 (4)
Fogginess in head (Psychiatric disorders) | 3 (4)
Headache (General disorders) | 13 (28)
Heart Racing (Cardiac disorders) | 8 (15)
Heavy limbs (Musculoskeletal and connective tissue disorders) | 5 (6)
Heavy head (General disorders) | 4 (7)
Insomnia (General disorders) | 3 (4)
Jaw Clenching (Musculoskeletal and connective tissue disorders) | 5 (8)
Jittery (General disorders) | 13 (33)
Lightheaded (General disorders) | 8 (22)
Limb Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (17)
Restlessness (General disorders) | 4 (5)
Stomach Ache (Gastrointestinal disorders) | 7 (10)
Stomach discomfort (Gastrointestinal disorders) | 6 (7)
Sweaty (General disorders) | 2 (4)
Tingling (General disorders) | 2 (3)
Tingling in hands (General disorders) | 2 (5)
Tingling in Head (General disorders) | 2 (2)
Tired (General disorders) | 8 (11)
Unfocused (Psychiatric disorders) | 9 (16)
Head Pressure (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No